CLINICAL TRIAL: NCT03282370
Title: Evaluate the Safety and Immunogenicity of a Vero Cell - Derived Inactivated Japanese Encephalitis Vaccine (JECEVAX) Produced by VABIOTECH (Vietnam) in Vietnamese Children Aged 9-24 Months
Brief Title: Evaluate Safety and Immunogenicity of a Vero Cell-Derived JE Vaccine in 9-24 Months of Age Children in Vietnam
Acronym: JECEVAX-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Ministry of Science and Technology, Vietnam (Other Government); Ministry of Health, Vietnam (Other Government)
Responsible Party: Principal Investigator, Vu Dinh Thiem, Head, Department of Epidemiology, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-JECEVAX-3
Record Dates: First submitted 2017-07-01; First posted 2017-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; JECEVAX; Vietnam
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JECEVAX (Experimental): JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.5 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 28-34 days
  Interventions: Biological: JECEVAX
- JEVAX (Active Comparator): JEVAX - VABIOTECH Vietnam Liquid form Composition: 1,0 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 28-34 days
  Interventions: Biological: JEVAX

INTERVENTIONS:
Biological: JEVAX — JEVAX - VABIOTECH Vietnam Liquid form Subcutaneous injection 0.5ml/dose, 2 doses, 28-34 days interval
  Arms: JEVAX
Biological: JECEVAX — JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.5 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 28-34 days
  Arms: JECEVAX

SUMMARY:
A study of the study vaccine (JECEVAX- VABIOTECH-Vietnam) and a licensed vaccine (JEVAX-VABIOTECH-Vietnam) is conducted in Vietnamese children, aged 9 to 24 months to assess the safety of the study vaccine compares to licenced vaccine. Two hundred and twenty children are enrolled and randomly assigned into 2 groups (110 children/group), each of which receive 2 doses of study / control vaccine subcutaneously, at 28-34 days interval. Safety data included immediate reaction at the injection site and systemic reaction within 30 min of administration, solicited and unsolicited adverse events occurs from the 1st dose to 28-34 days after first dose and from the second dose to 28-34 days after 2nd dose. SAE (from start of first dose to 28-34 days after second dose).

DETAILED DESCRIPTION:
Mouse brain-derived Japanese Encephalitis (JE) vaccine was developed in Vietnam since 1989 with the support from WHO and BIKEN institute, Japan. It helped Viet Nam prevents Japanese Encephalitis outbreaks successfully during those years.

However, mouse brain-derived JE vaccine production requires companies to compliance various requirements from WHO. Especially, WHO has a plan to replace the mouse brain-derived JE vaccines with Cell culture-derived JE vaccines.

Vero cell-derived vaccine technology shows many advantages compares to Mouse brain-derived vaccine technology. VABIOTECH has been approved and sponsored by the Ministry of Science and Technology to produce Vero cell - derived JE vaccine. The vaccine demonstrated a good safety and immunogenicity profile in animal models. The vaccine has been proven safety in volunteer adults and in phase 2 which evaluated the safety and immunogenicity of 3 difference antigen concentrations.

In this study, a selected dose of the studied vaccine (JECEVAX) derived from phase 2 will be compared the safety with a licensed vaccine (JEVAX-VABIOTECH Vietnam) in Vietnamese children, aged 9-24 months to assess the safety and immunogenicity. Two hundred and twenty children are enrolled and randomly assigned into 2 groups (110 children/group), each of which receive 2 doses of investigate vaccines or control vaccine subcutaneously, at 28-34 days interval. Safety data included immediate reaction at the injection site and systemic reaction within 30 min of administration, solicited and unsolicited adverse events occurs from the 1st dose to 28-34 days after first dose (up to date of 2nd dose) and from the second dose to 28-34 days after 2nd dose (up to date of 3rd visit). SAE (from start of first dose to 28-34 days after second dose - date of 3rd visit).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children of both sexes, 9-24 months of age;
* Have not been vaccinated with JE vaccine;
* Parents/legally guardians agree their children to participate in the study and sign the paper informed consent.

Exclusion Criteria:

* Currently has chronic diseases (cardiovascular, liver and spleen related etc);
* Currently has acute diseases;
* Use of immunocompromised treatment within 4 weeks of enrollment;
* Being immunocompromised and autoimmune diseases (HIV, lupus);
* The family history of immunocompromised;
* History of febrile seizure;
* Allergic to any vaccine component;
* Fever (>38 Celsius degree) within 3 days before vaccination or at enrollment;
* Malnourished (2nd grade or above);
* Blood disorder;
* Use of vaccines which have not been licenced 7 days before enrolment in this study

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 655 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-04-08 (Actual)

PRIMARY OUTCOMES:
Percent of participants with treatment-related adverse events during study period. | Up to 28-34 days after 2nd dose
  Percent of participants with solicited and unsolicited adverse events after each dose of vaccine: immediately injection site and systemic AEs after vaccination (within 30 min), solicited AEs within 7 days after each dose, unsolicited AEs from date 1st dose 1 to date of dose 2 and from date of 2nd dose to 28-34 day post 2nd dose (3rd visit), as assessed by CTCAE v.4.0.
Percent of participants who has antibody sero-conversion in study group and control group at 28-34 days post dose 2. | Up to 28-34 days after 2nd dose
  Serum samples will be taken before 1 dose and 28-34 days post 2nd dose to be tested for JE antibody by PRNT.

SECONDARY OUTCOMES:
Frequencies of participants with treatment-related SAE during study period | Up to 28-34 days after the 2nd dose (3rd visit)
  Frequencies of participants with treatment-related SAE during study period of JECEVAX compared to that of JEVAX, as assessed by CTCAE ver 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Thiem D Vu, MD., PhD., Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (4):
- Vietnam (4):
  - Hoa Binh Provincial Preventive Medicine Center, Hòa Bình, Hoa Binh
  - Hoa Binh City Health Center, Hòa Bình, Hoa Binh
  - District Health Center, Thanh Sơn, Phu Tho
  - Phu Tho Preventive Medicine Center, Việt Trì, Phu Tho

IPD SHARING:
Plan to Share IPD: No
Individual data with identification removed are to be available for Ethical committee, Ministry of Health and National Foundation of Science and Technology Development to avoid misuse of data.
  Public shared data will be in the form of summarised tables and figures.